CLINICAL TRIAL: NCT00095433
Title: An Extension Study to Evaluate the Safety and Tolerability of Multiple-Dose Intravitreal Injections of rhuFab V2 in Subjects With Neovascular Age-Related Macular Degeneration Who Have Completed the Treatment Phase of a Genentech-Sponsored Phase I or Phase I/II rhuFab V2 Study
Brief Title: Extension Study of rhuFab V2 in Subjects With Neovascular Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Masking: None | Purpose: Treatment
Other Study IDs: FVF2508g
Record Dates: First submitted 2004-11-04; First posted 2004-11-05 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Macular Degeneration
Keywords: AMD; Neovascular age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 (ranibizumab)

SUMMARY:
This is a Phase III, open-label, multicenter extension study of intravitreally administered ranibizumab in subjects with primary or recurrent subfoveal choroidal neovascularization (CNV) secondary to AMD who have completed the treatment phase of a Genentech sponsored Phase I or Phase I/II ranibizumab protocol (FVF1770g, FVF2128g, or FVF2425g).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age >=50 years
* Completion of the treatment phase of a Genentech sponsored Phase I or I/II ranibizumab protocol (FVF1770g, FVF2128g, or FVF2425g)

Exclusion Criteria:

* CNV in either eye due to other causes such as ocular histoplasmosis, trauma, or pathologic myopia
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* Subretinal hemorrhage in the study eye that involves the fovea, if the size of the hemorrhage is either >=50% of the total lesion area or >=1 DA in size
* Intraocular surgery (including cataract surgery) in the study eye within 1 month preceding Week 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >=30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* Laser photocoagulation (subfoveal, juxtafoveal, or extrafoveal) in the study eye within 30 days preceding Week 0
* Prior treatment with external-beam radiation therapy or transpupillary thermotherapy (TTT) in the study eye
* Previous treatment with verteporfin in the study eye within 30 days preceding Week 0
* Treatment with verteporfin in the non-study eye within 7 days preceding Week 0
* History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye
* Previous participation in a clinical trial (for either eye) involving antiangiogenic drugs other than ranibizumab (e.g., pegaptanib, anecortave acetate, protein kinase C inhibitors, etc.)
* Previous participation in any studies of investigational drugs within 1 month preceding Week 0 (excluding vitamins and minerals studies)
* Discontinuation from a ranibizumab study due to an adverse event judged by the investigator to be possibly or probably related to ranibizumab
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications
* Inability to comply with study or follow up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)